CLINICAL TRIAL: NCT03635957
Title: A Multicenter, Efficacy and Safety Study of Methotrexate to Increase Response Rates in Patients With Uncontrolled Gout Receiving KRYSTEXXA® (Pegloticase) (MIRROR Open-Label [OL])
Brief Title: Study of Pegloticase (KRYSTEXXA®) Plus Methotrexate in Patients With Uncontrolled Gout
Acronym: MIRROR OL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-KRY-201
Record Dates: First submitted 2018-08-09; First posted 2018-08-17 (Actual); Results first posted 2020-11-18 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Gout
Keywords: gout; uncontrolled gout
MeSH Terms: conditions — Gout | interventions — Pegloticase; Methotrexate; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pegloticase With Methotrexate (MTX) (Experimental): Run-In Period: oral MTX at a dose of 15 mg weekly for 4 weeks prior to the first dose of pegloticase.
  Pegloticase + Immunomodulator (IMM) Period: pegloticase 8 mg administered intravenously (IV) every 2 weeks from Day 1 through the Week 50 Visit for a total of 26 infusions. MTX 15 mg weekly on the same day each week, within 1 to 3 days prior to each pegloticase infusion and one additional weekly dose after the last infusion.
  Interventions: Biological: Pegloticase; Drug: Methotrexate (MTX); Drug: Standard Gout Flare Prophylaxis; Drug: Infusion Reaction (IR) Prophylaxis; Dietary Supplement: Folic Acid

INTERVENTIONS:
Biological: Pegloticase — pegloticase administered intravenously (IV)
Drug: Methotrexate (MTX) — oral MTX
Drug: Standard Gout Flare Prophylaxis — It is required that before a subject begins the Pegloticase + IMM Period, he or she has been taking at least one protocol standard gout flare prophylaxis regimen (i.e. colchicine and/or nonsteroidal anti-inflammatory drugs and/or low-dose prednisone ≤10 mg/day) for ≥1 week before the first dose of pegloticase and continues flare prophylaxis per American College of Rheumatology guidelines [Khanna D et al.2012] for the greater of 1) 6 months, 2) 3 months after achieving target serum urate (sUA < 6 mg/dL) for patients with no tophi detected on physical exam, or 3) 6 months after achieving target serum urate (sUA < 5 mg/dL) for patients with one or more tophi detected on initial physical exam that have since resolved.
Drug: Infusion Reaction (IR) Prophylaxis — For IR prophylaxis, fexofenadine (60 mg or 180 mg orally based on the Principal Investigator's discretion) will be taken the day before each infusion; fexofenadine (60 mg or 180 mg orally based on the Principal Investigator's discretion) and acetaminophen (1000 mg orally) will be taken the morning of each infusion; and methylprednisolone (125 mg IV) given over the infusion duration 10-30 minutes (recommended) or hydrocortisone (200 mg IV) will be administered immediately prior to each infusion.
Dietary Supplement: Folic Acid — Subjects will also take folic acid 1 mg orally every day beginning at Week -4 (the start of MTX) and continuing until prior to the Week 52 Visit.

SUMMARY:
The overall objective of the study is to assess the efficacy, safety, tolerability, and pharmacokinetics (PK) of the concomitant use of pegloticase with methotrexate (MTX) to enhance the response rate seen with pegloticase alone in adults with uncontrolled gout.

DETAILED DESCRIPTION:
The study design will include: 1) up to a 2-week Screening Period (screening should be complete within 2 weeks prior to Week -4), 2) a 4-week MTX Run in Period (Week - 4 through Day 1); 3) a 52-week Pegloticase + IMM (immunomodulator), (Pegloticase + MTX) Period 4) a Safety Follow-up (Phone/Email/Site Visit) and 5) a 3 and 6 month Post Treatment Follow-up.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent.
2. Willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the study.
3. Adult men or women ≥18 to ≤65 years of age.
4. Women of childbearing potential (including those with an onset of menopause <2 years prior to screening, non-therapy-induced amenorrhea for <12 months prior to screening, or not surgically sterile [absence of ovaries and/or uterus]) must have negative serum/urine pregnancy tests during the Screening/(methotrexate) MTX Run in Period; participants must agree to use 2 reliable forms of contraception during the study, one of which is recommended to be hormonal, such as an oral contraceptive. Hormonal contraception must be started ≥1 full cycle prior to Week -4 (start of MTX dosing) and continue for 30 days after the last dose of pegloticase or at least one ovulatory cycle after the last dose of MTX (whichever is the longest duration after the last dose of pegloticase or MTX). Highly effective contraceptive methods (with a failure rate <1% per year), when used consistently and correctly, include implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence, or vasectomized partner.
5. Men who are not vasectomized must not impregnant their female partner during the study and for at least 3 months after the last dose of MTX.
6. Hyperuricemia at the Screening, Week -4, or Week -2 Visit of the Screening/MTX Run in Period, as documented by sUA ≥6 mg/dL.
7. Uncontrolled gout, defined as meeting the following criteria:

   serum uric acid (sUA) ≥6 mg/dL prior to entry into the pegloticase +IMM Period (any laboratory tests during screening up to and including during the MTX Run in Period) and at least 1 of the following: inability to maintain sUA <6 mg/dL on other urate-lowering therapy; intolerable side effects associated with current urate-lowering therapy; functionally limiting tophaceous deposits (including those detected clinically or by dual-energy computed tomography [DECT] imaging)
8. Able to tolerate MTX 15 mg for 4 weeks during the MTX Run-in Period prior to the first dose of pegloticase.

Exclusion Criteria:

1. Weight >160 kg (352 pounds).
2. Any serious acute bacterial infection, unless treated and completely resolved with antibiotics at least 2 weeks prior to the Week -4 Visit of the MTX Run-in Period.
3. Severe chronic or recurrent bacterial infections, such as recurrent pneumonia or chronic bronchiectasis.
4. Current immunocompromised condition, including current or chronic treatment with systemic immunosuppressive agents, including prednisone >10 mg/day or equivalent dose of other corticosteroid.
5. History of any transplant surgery requiring maintenance immunosuppressive therapy.
6. Known history of hepatitis B virus surface antigen positivity or hepatitis B DNA positivity.
7. Known history of hepatitis C virus RNA positivity.
8. Human immunodeficiency virus (HIV) positivity (tested at the Screening Visit).
9. Glucose-6-phosphate dehydrogenase (G6PD) deficiency (tested at the Screening Visit).
10. Severe chronic renal impairment (glomerular filtration rate <25 mL/min/1.73 m^2) or currently on dialysis.
11. Non-compensated congestive heart failure or hospitalization for congestive heart failure within 3 months of the Screening Visit, uncontrolled arrhythmia, treatment for acute coronary syndrome (myocardial infarction or unstable angina), or uncontrolled blood pressure (>160/100 mmHg) at the end of the Screening/MTX Run-in Period.
12. Pregnant, planning to become pregnant, breastfeeding, planning to impregnant female partner, or not on an effective form of birth control, as determined by the Investigator.
13. Prior treatment with pegloticase (KRYSTEXXA®), another recombinant uricase (rasburicase), or concomitant therapy with a polyethylene glycol-conjugated drug.
14. Known allergy to pegylated products or history of anaphylactic reaction to a recombinant protein or porcine product.
15. Contraindication to MTX treatment or MTX treatment considered inappropriate.
16. Known intolerance to MTX.
17. Receipt of an investigational drug within 4 weeks or 5 half-lives, whichever is longer, prior to MTX administration at Week -4 or plans to take an investigational drug during the study.
18. Current liver disease, as determined by alanine transaminase or aspartate transaminase levels >3 times upper limit of normal at the Screening Visit.
19. Currently receiving systemic or radiologic treatment for ongoing cancer, excluding non melanoma skin cancer.
20. History of malignancy within 5 years other than non-melanoma skin cancer or in situ carcinoma of cervix.
21. Uncontrolled hyperglycemia with a plasma glucose value >240 mg/dL at screening that is not subsequently controlled by the end of the Screening/MTX Run-in Period.
22. Diagnosis of osteomyelitis.
23. Known history of hypoxanthine-guanine phosphoribosyl-transferase deficiency, such as Lesch-Nyhan and Kelley-Seegmiller syndrome.
24. Unsuitable candidate for the study, based on the opinion of the Investigator (e.g., cognitive impairment), such that participation might create undue risk to the participant or interfere with the participant's ability to comply with the protocol requirements or complete the study.
25. Alcohol use in excess of 3 alcoholic beverages per week.
26. Currently receiving allopurinol and unable to discontinue medication 7 days prior to MTX dosing at Week -4 and unable to discontinue treatment during the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2020-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (6):
- United States (6):
  - Orthopedic Physicians Alaska, Anchorage, Alaska
  - Arizona Arthritis & Rheumatology -West Valley, Glendale, Arizona
  - Arizona Arthritis & Rheumatology -East Valley, Mesa, Arizona
  - Avail Clinical Research, DeLand, Florida
  - Western Washington Arthritis Clinic, Bothell, Washington
  - Arthritis Northwest PLLC, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Botson JK, Obermeyer K, LaMoreaux B, Zhao L, Weinblatt ME, Peterson J. Improved joint and patient-reported health assessments with pegloticase plus methotrexate co-therapy in patients with uncontrolled gout: 12-month exploratory outcomes of the MIRROR open-label trial. Arthritis Res Ther. 2022 Dec 27;24(1):281. doi: 10.1186/s13075-022-02979-4. PMID 36575505
- [Derived] Botson JK, Tesser JRP, Bennett R, Kenney HM, Peloso PM, Obermeyer K, Song Y, LaMoreaux B, Zhao L, Xin Y, Chamberlain J, Ramanathan S, Weinblatt ME, Peterson J. A multicentre, efficacy and safety study of methotrexate to increase response rates in patients with uncontrolled gout receiving pegloticase (MIRROR): 12-month efficacy, safety, immunogenicity, and pharmacokinetic findings during long-term extension of an open-label study. Arthritis Res Ther. 2022 Aug 25;24(1):208. doi: 10.1186/s13075-022-02865-z. PMID 36008814
- [Derived] Dalbeth N, Becce F, Botson JK, Zhao L, Kumar A. Dual-energy CT assessment of rapid monosodium urate depletion and bone erosion remodelling during pegloticase plus methotrexate co-therapy. Rheumatology (Oxford). 2022 Nov 28;61(12):4898-4904. doi: 10.1093/rheumatology/keac173. PMID 35293984
- [Derived] Botson JK, Tesser JRP, Bennett R, Kenney HM, Peloso PM, Obermeyer K, LaMoreaux B, Weinblatt ME, Peterson J. Pegloticase in Combination With Methotrexate in Patients With Uncontrolled Gout: A Multicenter, Open-label Study (MIRROR). J Rheumatol. 2021 May;48(5):767-774. doi: 10.3899/jrheum.200460. Epub 2020 Sep 15. PMID 32934137

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was dosed with methotrexate (MTX) in the Run-In Period (MTX tolerance period) but was lost to follow up prior to the per protocol enrollment at Day 1. This participant was a screen failure but is included in the Run-in period data (including safety).
Groups:
- All Participants: Run-In Period: oral MTX at a dose of 15 mg weekly for 4 weeks prior to the first dose of pegloticase.
  Pegloticase + Immunomodulator (IMM) Period: pegloticase 8 mg administered intravenously (IV) every 2 weeks from Day 1 through the Week 50 Visit for a total of 26 infusions. MTX 15 mg weekly on the same day each week, within 1 to 3 days prior to each pegloticase infusion and one additional weekly dose after the last infusion.
Period: Run-In Period
Arm/Group | All Participants
Started | 15
Completed | 14
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Pegloticase + IMM Period
Arm/Group | All Participants
Started | 14
Completed Study at 24 Weeks-Amendment 1 | 1
Completed Study at 52 Weeks-Amendment 2 | 10
Discontinued Study Treatment Early | 5
Had 3-Month Follow-up | 7
Had 6-Month Follow-up | 6
Completed (1 participant completed study under Amend. 1 at Week 24. Amend. 2 extended the study to 52 weeks.) | 11
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Population: Modified intention-to-treat (mITT) population: all enrolled participants who received ≥1 dose of pegloticase.
Groups:
- Pegloticase With Methotrexate (MTX): Run-In Period: oral MTX at a dose of 15 mg weekly for 4 weeks prior to the first dose of pegloticase.
  Pegloticase + IMM Period: pegloticase 8 mg administered IV every 2 weeks from Day 1 through the Week 50 Visit for a total of 26 infusions. MTX 15 mg weekly on the same day each week, within 1 to 3 days prior to each pegloticase infusion and one additional weekly dose after the last infusion.
Arm/Group | Pegloticase With Methotrexate (MTX)
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (8.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Serum Uric Acid (sUA) [Mean (Standard Deviation); unit: mg/dL] — Baseline is defined as the last measurement taken prior to the first infusion of pegloticase in the pegloticase + IMM period.
  mg/dL | 9.16 (2.486)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Serum Uric Acid (sUA < 6 mg/dL) Responders During Month 6
Description: Serum uric acid (sUA < 6 mg/dL) responders are defined as participants achieving and maintaining sUA < 6 mg/dL for at least 80% of the time during Month 6 (Weeks 20, 22, and 24). Month 6 includes pre-infusion and post-infusion sUA assessments at Week 20, pre-infusion and post-infusion sUA assessments at Week 22, pre-infusion assessments at Week 24, and unscheduled sUA assessments between Week 20 and Week 24.
Time Frame: Month 6 (Weeks 20, 22, and 24)
Population: Modified Intent to Treat Population: all enrolled participants who received at least 1 dose of pegloticase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegloticase With Methotrexate (MTX)
Number analyzed (Participants) | 14
percentage of participants | 78.6 [49.2 to 95.3]

2. Secondary Outcome: Percentage of Serum Uric Acid (sUA < 6 mg/dL) Responders During Month 3
Description: Serum uric acid (sUA < 6 mg/dL) responders are defined as participants achieving and maintaining sUA < 6 mg/dL for at least 80% of the time during Month 3 (Weeks 10, 12, and 14). Month 3 includes pre-infusion and post-infusion sUA assessments at Week 10, pre-infusion and post-infusion sUA assessments at Week 12, pre-infusion assessments at Week 14, and unscheduled assessments between Week 10 and Week 14 pre-infusion.
Time Frame: Month 3 (Weeks 10, 12, and 14)
Population: Modified Intent to Treat Population: all enrolled participants who received at least 1 dose of pegloticase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegloticase With Methotrexate (MTX)
Number analyzed (Participants) | 14
percentage of participants | 78.6 [49.2 to 95.3]

3. Secondary Outcome: Percentage of Serum Uric Acid (sUA < 6 mg/dL) Overall Responders
Description: Serum uric acid (sUA < 6 mg/dL) overall responders are defined as participants achieving and maintaining sUA < 6 mg/dL for at least 80% of the time during Month 3 and Month 6 (Weeks 10, 12, 14, 20, 22, and 24) combined. Participants with more than one sUA result in Month 3 and Month 6 are considered responders if a participant's weighted proportion of hours that sUA is < 6 mg/dL is greater than or equal to 80%. Participants with the proportion of hours less than 80% are counted as non-responders. Participants with only one value in Month 3 and Month 6 are considered overall responders if they are considered responders in both Month 3 and Month 6.
Time Frame: Month 3 and Month 6 combined (Weeks 10, 12, 14, 20, 22, and 24)
Population: Modified Intent to Treat Population: all enrolled participants who received at least 1 dose of pegloticase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegloticase With Methotrexate (MTX)
Number analyzed (Participants) | 14
percentage of participants | 78.6 [49.2 to 95.3]

4. Secondary Outcome: Percentage of Serum Uric Acid (sUA < 5 mg/dL) Responders During Month 3
Description: Serum uric acid (sUA < 5 mg/dL) responders are defined as participants achieving and maintaining sUA < 5 mg/dL for at least 80% of the time during Month 3. Month 3 includes pre-infusion and post-infusion sUA assessments at Week 10, pre-infusion and post-infusion sUA assessments at Week 12, pre-infusion assessments at Week 14, and unscheduled assessments between Week 10 and Week 14 pre-infusion.
Time Frame: Month 3 (Weeks 10, 12, and 14)
Population: Modified Intent to Treat Population: all enrolled participants who received at least 1 dose of pegloticase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegloticase With Methotrexate (MTX)
Number analyzed (Participants) | 14
percentage of participants | 78.6 [49.2 to 95.3]

5. Secondary Outcome: Percentage of Serum Uric Acid (sUA < 5 mg/dL) Responders During Month 6
Description: Serum uric acid (sUA < 5 mg/dL) responders are defined as participants achieving and maintaining sUA < 5 mg/dL for at least 80% of the time during Month 6. Month 6 includes pre-infusion and post-infusion sUA assessments at Week 20, pre-infusion and post-infusion sUA assessments at Week 22, pre-infusion assessments at Week 24, and unscheduled sUA assessments between Week 20 and Week 24.
Time Frame: Month 6 (Weeks 20, 22, and 24)
Population: Modified Intent to Treat Population: all enrolled participants who received at least 1 dose of pegloticase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegloticase With Methotrexate (MTX)
Number analyzed (Participants) | 14
percentage of participants | 78.6 [49.2 to 95.3]

6. Secondary Outcome: Percentage of Serum Uric Acid (sUA < 5 mg/dL) Overall Responders
Description: Serum uric acid (sUA < 5 mg/dL) overall responders are defined as participants achieving and maintaining sUA < 5 mg/dL for at least 80% of the time during Month 3 and Month 6 (Weeks 10, 12, 14, 20, 22, and 24) combined. Participants with more than one sUA result in Month 3 and Month 6 are considered responders if a participant's weighted proportion of hours that sUA is < 6 mg/dL is greater than or equal to 80%. Participants with the proportion of hours less than 80% are counted as non-responders. Participants with only one value in Month 3 and Month 6 are considered overall responders if they are considered responders in both Month 3 and Month 6.
Time Frame: Month 3 and Month 6 combined (Weeks 10, 12, 14, 20, 22, and 24)
Population: Modified Intent to Treat Population: all enrolled participants who received at least 1 dose of pegloticase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pegloticase With Methotrexate (MTX)
Number analyzed (Participants) | 14
percentage of participants | 78.6 [49.2 to 95.3]

7. Secondary Outcome: Mean Change in sUA From Pegloticase Baseline to Weeks 14, 24, 36, 52
Description: The mean change from baseline is based on observed values in participants remaining on treatment at given time point. For sUA values less than the lower limit of detection (up to 1.5 mg/dL), 0 is used in the analysis.
Time Frame: Baseline (defined as the last measurement taken prior to the first infusion of pegloticase in the pegloticase + IMM period), Pre- and Post-Infusion at Weeks 14, 24, 36 and Week 52
Population: Modified Intent to Treat Population: all enrolled participants who received at least 1 dose of pegloticase. Participants with a measurement at given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pegloticase With Methotrexate (MTX)
Number analyzed (Participants) | 14
mg/dL
  Change at Week 14 - pre-infusion: number analyzed (Participants) | 11
  Change at Week 14 - pre-infusion | -9.27 (2.810)
  Change at Week 14 - post-infusion: number analyzed (Participants) | 10
  Change at Week 14 - post-infusion | -9.31 (2.959)
  Change at Week 24 - pre-infusion: number analyzed (Participants) | 11
  Change at Week 24 - pre-infusion | -9.27 (2.810)
  Change at Week 24 - post-infusion: number analyzed (Participants) | 5
  Change at Week 24 - post-infusion | -9.48 (4.135)
  Change at Week 36 - pre-infusion: number analyzed (Participants) | 10
  Change at Week 36 - pre-infusion | -8.13 (3.975)
  Change at Week 36 - post-infusion: number analyzed (Participants) | 8
  Change at Week 36 - post-infusion | -9.41 (3.293)
  Change at Week 52: number analyzed (Participants) | 10
  Change at Week 52 | -8.15 (4.086)

ADVERSE EVENTS:
Time Frame: From first dose of study drug through the end of treatment plus 30 days. Mean duration of MTX Treatment during the MTX Run-in Period was 23.0 days, and during the Pegloticase+IMM Period was 242.4 days. Mean duration of pegloticase treatment during the Pegloticase + IMM Period was 242.4 days.
Description: Treatment-emergent adverse events (TEAEs) are presented. The Intent to Treat population (all enrolled participants who took at least one dose of MTX) is used to present TEAEs for the run-in period. Modified Intent to Treat Population (all enrolled participants who received at least 1 dose of pegloticase) is used to present TEAEs for the Pegloticase + IMM Period.
Groups:
- Run-In Period: MTX: Run-In Period: oral MTX at a dose of 15 mg weekly for 4 weeks prior to the first dose of pegloticase.
- Pegloticase + IMM Period: Pegloticase + MTX: Pegloticase + IMM Period: pegloticase 8 mg administered IV every 2 weeks from Day 1 through the Week 50 Visit for a total of 26 infusions. MTX 15 mg weekly on the same day each week, within 1 to 3 days prior to each pegloticase infusion and one additional weekly dose after the last infusion.
Arm/Group | Run-In Period: MTX | Pegloticase + IMM Period: Pegloticase + MTX
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/14
Other Adverse Events (participants affected / at risk) | 10/15 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In Period: MTX (N=15) | Pegloticase + IMM Period: Pegloticase + MTX (N=14)
Bacterial Sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In Period: MTX (N=15) | Pegloticase + IMM Period: Pegloticase + MTX (N=14)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Dry Eye (Eye disorders) | 1 | 0
Eye Irritation (Eye disorders) | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Tooth Impacted (Gastrointestinal disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Chronic Sinusitis (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 3
Carbuncle (Infections and infestations) | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 3
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 3
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Liver Function Test Increased (Investigations) | 0 | 1
Gout (Metabolism and nutrition disorders) | 5 | 13
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Parosmia (Nervous system disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
One participant was dosed with MTX in the Run-In Period (MTX tolerance period) but was lost to follow up prior to the per protocol enrollment at Day 1. This participant was a screen failure but is included in Run-in period data (including safety).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any Investigator/institution that plans on presenting or publishing results provide written notification of their request a minimum of 60 days prior to presentation or publication. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsors' Intellectual Property rights.

DOCUMENTS (2):
  • Study Protocol (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT03635957/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT03635957/SAP_001.pdf